CLINICAL TRIAL: NCT03998241
Title: Joint Position Sense in Individuals With Anterior Knee Pain
Status: Completed | Type: Observational
Sponsor: University of Stellenbosch (Other)
Collaborators: National Research Foundation of South Africa (Other)
Responsible Party: Principal Investigator, Dominique Leibbrandt, Dr Dominique Leibbrandt (PhD Physiotherapy), Postdoctoral Researcher in Faculty of Health and Rehabilitation Sciences, University of Stellenbosch
Other Study IDs: DLeibbrandt
Record Dates: First submitted 2019-06-06; First posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Anterior Knee Pain Syndrome; Proprioceptive Disorders
Keywords: patellofemoral pain; joint position sense; movement analysis
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Somatosensory Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention was provided — No intervention given
  Other Names: None given

SUMMARY:
Introduction Anterior knee pain (AKP) commonly affects physically active as well as sedentary individuals and the aetiology remains unknown. Altered joint position sense (JPS) impacts accurate motor action and knee joint stability. It is unclear whether people with AKP have altered JPS. The aim of this study was to investigate the JPS of individuals with AKP.

Methods A descriptive cross-sectional design was used to measure JPS in twenty-five participants with unilateral or bilateral AKP. The Vicon 3D motion analysis system was used to assess JPS by means of active joint position sense testing during single leg squat and active knee extension in sitting. Target angles were self-determined based on each participant's capabilities. The absolute error (AE) was used as the main outcome measure. Impaired JPS was classified as an AE equal to or greater than five degrees.

DETAILED DESCRIPTION:
Research Design CAF Human motion analysis Unit, Faculty of Medicine and Health Sciences, Stellenbosch University. Ethical approval was obtained from the Health Research Ethics Committee of Stellenbosch University under reference number S16/10/197. This study was conducted as part of a master's thesis project (Rhode 2018).

Sampling and Recruitment Sample recruitment was aimed to attract individuals with AKP from different socio-economic backgrounds, sporting codes and areas. Letters of invitation were sent to various universities, sports clinics, physiotherapy practices and sporting clubs.

Study Procedure Measurement Tools Vicon 3D motion analysis system The eight-camera Vicon T-20-series motion analysis system (Vicon Motion Systems Ltd., Oxford, UK) with Nexus 1.7 software was used to assess joint position sense (JPS). The Vicon has demonstrated high accuracy and reliability and has been shown to have less than a 1.5-degree error (Ehara et al 1997). Retro-reflective markers with a diameter of 9.5mm were used. Dynamic calibration was performed according to standard laboratory protocol, and the Vicon T-wand was placed on a 3D Bertec force plate (Bertec Corporation Ltd.), which is synchronized with the Vicon motion analysis system.

H-Frame An H-frame was constructed based on a study by Clark et al (2016). The function of the H-frame was that of a range of motion (ROM) guide when establishing the target angle (TA) for participants during the test trial. The H-frame was positioned so that the rubber band (crossbar) makes contact with the distal part of the patella during single leg squat (SLS) and that the crossbar touches the skin overlying the anterior ankle joint line during active knee extension (AKE). The H-frame was removed during the test procedure.

Kujala/anterior knee pain scale (AKPS) questionnaire The AKPS is a 13-item knee functional questionnaire. This scale is scored out of 100, with a higher score indicating less disability. The AKPS demonstrated high reliability and responsiveness in a population of patients with AKP (Watson et al 2005).

Visual analogue pain scale (VAS) This VAS scale is a well-known outcome measure to evaluate levels/intensity of pain (Crossley et al 2016). The VAS is scored from 0 (no pain) to 10 (maximum pain). The VAS demonstrates good reliability and responsiveness among a population of patients with AKP (Green et al 2014).

Lower extremity functional scale (LEFS) questionnaire The LEFS consists of 20 items that measure the ability to perform various functional activities and activities of daily life. The LEFS is scored out of a maximum score of 80. The LEFS demonstrates high reliability and responsiveness in the population of patients with AKP (Watson et al 2005).

Criteria for positive and negative knee joint position sense The main outcome measurements for knee JPS testing was absolute error (AE). AE refers to the difference between the test or target angle and the reproduced angle. Absolute error represents accuracy without directional bias. For the purpose of this study, abnormal JPS was defined as an AE equal or greater than five degrees. This criterion was based on published research by Relph and Callaghan (2016) and Clark et al (2016) using healthy pain free participants. The mean AE from five trails for each test was used for statistical analysis (Selfe et al 2006).

Testing Procedures Initial screening To verify that participants met the inclusion criteria they completed a screening questionnaire via email. Prior to JPS testing, participants completed the AKP scale questionnaire (AKPS) and the LEFS questionnaire. A data collection form was used to collect participant personal details and variables including age, gender, body length, episodes and duration of AKP, area of symptoms, type of treatment received for AKP and sport participation.

Physical examination and diagnosis The diagnostic checklist was completed, and the physical examination was performed to confirm a diagnosis of AKP and to exclude other knee pathologies prior to testing. The physical examination (P/E) was conducted by the primary researcher (CR), who is an experienced physiotherapist. Additionally, anthropometrics (weight, BMI, leg length) were measured for each participant. Data were captured as part of participant demographics to describe this population group/participants.

Preparation for Vicon testing Participants were dressed in short pants, were barefoot, with clean shaven legs with no lotion on legs to ensure effective marker placement. Thirty retro-reflective markers were placed on bony landmarks according to lower limb Plug-in Gait model (Clark et al 2016). Additional pelvic markers, a sacral wand, two extra shin markers and extra anterior and posterior thigh markers where added, to ensure joint position sense accuracy. The primary researcher (CR) performed the marker placement assisted by a research assistant. Reflective markers were placed in the standing position in preparation for SLS and re-applied with the participant in the seated position to ensure accurate positioning of markers placements for active knee extension. A static and dynamic calibration were performed in both test positions.

Pain measurement During the test trials the participants were asked to verbally indicate the severity of their anterior knee pain using the VAS pain scale. Pain severity was measured at the start and end of proprioceptive testing.

Proprioceptive Testing All participants were familiarized with the proprioceptive test procedure by means of explanation, demonstration and a practice opportunity. The participants were asked to resume the test position i.e. (i) standing or (ii) sitting. The target angle was determined by each participant according to his/her capabilities and comfort level, i.e. the target angle was unique to each participant.

Single leg squat (SLS) Starting position For the SLS the participant supported one hands on a chair for balance. The participant was standing on the tested leg, while the other leg was slightly flexed at the hip and knee in a position that was comfortable for the participant.

Instructions to participant The participant was asked to do a SLS and stop in the mid-range. The participant was asked to briefly hold this mid-range angle to position the H-frame indicating this angle as the target angle (TA).

Test trial The participant was cued to squat down till they felt the cross bar of the H-frame. The participant was instructed to hold the SLS for five seconds to establish and familiarize themselves with the target angle (TA). The test trial was repeated five times.

Test procedure The participant was blindfolded, and the H-frame was removed. The participant was instructed to perform a SLS, and to indicate when they had reached the TA by shouting STOP. This position indicated the relative error (RE) and was maintained for five seconds to record the data. Testing was repeated five times. This number of repetitions has been recommended for JPS testing in previous research (Selfe et al 2006). SLS was repeated on the knees without AKP for comparison.

Sitting: active knee extension (AKE) Starting position The participant was seated on an 800mm high bar stool, with both feet supported. Each participant was positioned with the popliteal fossa approximately 5cm from the edge of the chair. The participant's arms were crossed over their chests comfortably to avoid obstruction of the pelvic markers.

Instructions to participants The participant actively extended the knee through the range of 90 degrees knee flexion to 0 degrees knee extension; thereafter they had to stop in the mid-range position. The participant was asked to briefly hold this mid-range angle to position the H-frame indicating this position as the TA. The participant was verbally cued to resume the starting position.

Test trial The participant actively extended the knee from the starting position of 90 degrees knee flexion to the TA. The participants were verbally cued to hold this position for five seconds to establish the TA. Thereafter the participant was asked to return to the starting position of the knee in 90 degrees flexion. The test trail was repeated five times.

Testing The H-frame was removed at the commencement of AKE testing. The participant was asked to repeat AKE, indicating when the TA had been reached, by shouting STOP. This position indicated the relative error (RE) and the participants maintained this position for five seconds. Testing was repeated five times. The AKE was repeated on the knees without AKP for comparison.

Statistical Analyses All descriptive data (demographic information, functional and pain scales) were analyzed using descriptive statistics to indicate central tendencies in data (means and standard deviations). A non-pragmatic test approach was adopted by illustrating the ranges. Data was captured through the Vicon Nexus 3D motion analyses system. Chi-square calculations was performed to determine a significant difference in JPS between the knees with AKP and the knees without AKP during single leg stance and active knee extension.

ELIGIBILITY:
Inclusion Criteria:

Participants who adhered to the criteria listed below were considered for inclusion:

* Individuals aged between 14 and 40 years
* Insidious onset of clinical signs and symptoms of AKP (more than 3 months duration)
* Symptoms were provoked by prolonged sitting, squatting, stair-climbing and/or running.
* Participants needed to comply with the AKP screening tool and the diagnostic checklist (Leibbrandt & Louw 2017)

Exclusion Criteria:

Participants were excluded if they presented with the following:

* AKP had resulted from a traumatic event such as a motor vehicle accident
* Previous knee surgery or injuries
* Clinical evidence of other knee pathologies
* If they were experiencing any other lower extremity injuries

Ages: 14 Years to 40 Years | Sex: All
Age Groups: Child, Adult
Study Population: A total of 25 participants complied with the inclusion criteria (Table 1); with the majority being female (n=22). The participants had a mean age of 27.8 years and a mean BMI of 28.2 kg/m2 (range of 20.9- 45.7kg/m). Twelve (52%) of the participants reported having AKP symptoms in both knees and ten (40%) participants reported their right knee as most affected. Nineteen (76%) of the 25 participants reported being physically active and six (24%) were sedentary. The participants' mean usual pain level according to the VAS was 4.5/10.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Weight Bearing JPS during single leg squatting | Measured six times on the same day
  Active angle reproduction using Vicon movement analysis system
Non-weight bearing JPS during active knee extension | Measured six times on the same day
  Active angle reproduction using Vicon movement analysis system
Usual pain: Visual analogue scale (VAS) | Measured at recruitment (onset of research) and during testing procedures (active knee extension and single leg squatting)
  Visual analogue scale pain measurement ranging from 0 (no pain) to 10 (worst possible pain)
Anterior knee pain scale (AKPS) | Measured on the day of the assessment prior to motion analysis procedures
  Anterior knee pain specific scale to measure functional ability. Score is out of 100. a score of 100 indicates no functional impairment.
Lower extremity functional scale (LEFS) | Measured on the day of the assessment prior to motion analysis procedures
  A scale out of 80 to measure functional ability as a result of lower extremity injury. A score of 80 indicates no functional impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Stellenbosch Univeristy Medical Campus, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Relph N, Herrington L. The effects of knee direction, physical activity and age on knee joint position sense. Knee. 2016 Jun;23(3):393-8. doi: 10.1016/j.knee.2016.02.018. Epub 2016 Mar 21. PMID 27012638
- [Background] Ehara Y, Fujimoto H, Miyazaki S, Mochimaru M, Tanaka S, Yamamoto S (1997) Comparison of the performance of the 3D camera system II. Gait and Posture 5: 251-255
- [Background] Clark NC, Akins JS, Heebner NR, Sell TC, Abt JP, Lovalekar M, Lephart SM. Reliability and measurement precision of concentric-to-isometric and eccentric-to-isometric knee active joint position sense tests in uninjured physically active adults. Phys Ther Sport. 2016 Mar;18:38-45. doi: 10.1016/j.ptsp.2015.06.005. Epub 2015 Jun 18. PMID 26804382
- [Background] Watson CJ, Propps M, Ratner J, Zeigler DL, Horton P, Smith SS. Reliability and responsiveness of the lower extremity functional scale and the anterior knee pain scale in patients with anterior knee pain. J Orthop Sports Phys Ther. 2005 Mar;35(3):136-46. doi: 10.2519/jospt.2005.35.3.136. PMID 15839307
- [Background] Green A, Liles C, Rushton A, Kyte DG. Measurement properties of patient-reported outcome measures (PROMS) in Patellofemoral Pain Syndrome: a systematic review. Man Ther. 2014 Dec;19(6):517-26. doi: 10.1016/j.math.2014.05.013. Epub 2014 Jun 14. PMID 24997774
- [Background] Selfe J, Callaghan M, McHenry A, Richards J, Oldham J. An investigation into the effect of number of trials during proprioceptive testing in patients with patellofemoral pain syndrome. J Orthop Res. 2006 Jun;24(6):1218-24. doi: 10.1002/jor.20127. PMID 16705703
- [Result] Rhode C (2018). Proprioceptive differences in individuals with Anterior knee pain. Master's dissertation Stellenbosch: Stellenbosch University.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT03998241/Prot_SAP_000.pdf
  • Informed Consent Form (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT03998241/ICF_001.pdf